CLINICAL TRIAL: NCT00569166
Title: Paced Breathing for Hot Flashes: A Randomized Phase II Study
Brief Title: Three Different Programs of Paced Breathing in Treating Hot Flashes in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CDR0000579010; P30CA015083 (NIH); MC06C8 (Other: Mayo Clinic Cancer Center); 06-005157 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2007-12-05; First posted 2007-12-06 (Estimated); Results first posted 2011-12-06 (Estimated); Last update posted 2017-08-07 (Actual); Status verified 2011-11

CONDITIONS: Breast Cancer; Fatigue; Hot Flashes; Sleep Disorders
Keywords: fatigue; sleep disorders; ductal breast carcinoma in situ; lobular breast carcinoma in situ; breast cancer; hot flashes
MeSH Terms: conditions — Breast Neoplasms; Fatigue; Hot Flashes; Sleep Wake Disorders; Carcinoma, Intraductal, Noninfiltrating; Breast Carcinoma In Situ

STUDY DESIGN:
Who Masked: Investigator

ARMS (3):
- Paced breathing (15 min once daily, 6 breaths/min) (Active Comparator): Patients practice paced breathing for 15 minutes once daily, 6 breaths/min, 5-7 days weekly, following an instructional CD, for 8 weeks.
  Interventions: Behavioral: Paced breathing (15 min once daily, 6 breaths/min)
- Paced breathing (15 min twice daily, 6 breaths/min) (Active Comparator): Patients practice paced breathing for 15 minutes twice daily, 6 breaths/min, 5-7 days weekly, following an instructional CD, for 8 weeks.
  Interventions: Behavioral: Paced breathing (15 min twice daily, 6 breaths/min)
- Paced breathing (10 min once daily, 14 breaths/min) (Placebo Comparator): Patients practice paced breathing for 10 minutes once daily, 14 breaths /min, 5-7 days weekly, following an instructional CD, for 8 weeks.
  Interventions: Behavioral: Paced breathing (10 min once daily, 14 breaths/min)

INTERVENTIONS:
Behavioral: Paced breathing (15 min once daily, 6 breaths/min) — Patients practice paced breathing for 15 minutes once daily, 6 breaths/min, 5-7 days weekly, following an instructional CD, for 8 weeks.
  Arms: Paced breathing (15 min once daily, 6 breaths/min)
Behavioral: Paced breathing (15 min twice daily, 6 breaths/min) — Patients practice paced breathing for 15 minutes twice daily, 6 breaths/min, 5-7 days weekly, following an instructional CD, for 8 weeks.
  Arms: Paced breathing (15 min twice daily, 6 breaths/min)
Behavioral: Paced breathing (10 min once daily, 14 breaths/min) — Patients practice paced breathing for 10 minutes once daily, 14 breaths /min, 5-7 days weekly, following an instructional CD, for 8 weeks.
  Arms: Paced breathing (10 min once daily, 14 breaths/min)

SUMMARY:
RATIONALE: Paced breathing may be an effective way to reduce the number and severity of hot flashes in women who have survived breast cancer.

PURPOSE: This randomized phase II trial is comparing three different programs of paced breathing to see how well they work in treating hot flashes in women.

DETAILED DESCRIPTION:
OBJECTIVES:

* To assess feasibility and obtain initial estimates of efficacy of three different programs of paced breathing (15 minutes once a day at 6 breaths/minute vs 15 minutes twice a day at 6 breaths/minute vs 10 minutes once a day at 14 breaths/minute) on the frequency and severity of hot flashes in breast cancer survivors or patients not preferring to take hormones because of concern for breast cancer.
* To assess feasibility and obtain initial estimates of efficacy of three different programs of paced breathing on mood states, fatigue, sleep quality, and blood pressure measurement in breast cancer survivors or patients not preferring to take hormones because of concern for breast cancer.

OUTLINE: Patients are stratified by age (18-49 vs ≥ 50), frequency of hot flashes per day (< 4 vs 4-9 vs ≥ 10), and current tamoxifen, raloxifene, or aromatase inhibitor treatment (yes vs no). Patients are randomized to 1 of 3 treatment arms.

* Arm I: Patients practice paced breathing for 15 minutes once daily, 6 breaths/min, 5-7 days weekly, following an instructional compact disc (CD), for 8 weeks.
* Arm II: Patients practice paced breathing for 15 minutes twice daily, 6 breaths/min, 5-7 days weekly, following an instructional CD, for 8 weeks.
* Arm III: Patients practice paced breathing for 10 minutes once daily, 14 breaths /min, 5-7 days weekly, following an instructional CD, for 8 weeks.

All patients complete daily hot flash diaries, keep a blood pressure log, and complete the following questionnaires: Symptom Experience Diary, Profile of Mood States, Brief Fatigue Inventory, and Pittsburgh Sleep Quality Index.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* History of breast cancer including ductal carcinoma in situ or lobular carcinoma in situ

  - Treated with surgery and/or adjuvant therapy with a curative intent or patients not preferring to take hormones because of concern for breast cancer
* Frequent hot flashes (≥ 14 per week) of sufficient severity to make the patient desire treatment
* Presence of hot flashes for ≥ 1 month prior to study entry
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Pre- or post-menopausal
* Must possess a compact disc (CD) player
* Able to complete questionnaires alone or with assistance
* No active medical conditions preventing compliance with a practice of slow deep breathing including active asthma, chronic obstructive pulmonary disease, or congestive heart failure
* No uncontrolled hypertension (defined as systolic blood pressure (BP) ≥ 160 mm Hg and/or diastolic BP ≥ 100 mm Hg on 2 separate visits)

PRIOR CONCURRENT THERAPY:

* No current (within the past month) practice of yoga or breathing exercises
* No other concurrent agents for treating hot flashes (e.g., gabapentin, venlafaxine, paroxetine, citalopram, sertraline, natural products such as soy or sage supplements, flaxseed, or black cohosh)

  - Concurrent stable dose antidepressants started within the past 30 days allowed
* No concurrent hormonal agents and/or antineoplastic chemotherapy - Tamoxifen, raloxifene, and aromatase inhibitors are allowed if patient has been on a constant dose for ≥ 4 weeks and does not plan to stop the treatment during the course of the study

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2007-03; Primary Completion 2010-02 (Actual); Study Completion 2012-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amit Sood, MD, Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic Cancer Center, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One-hundred and five (105) participants were recruited at Mayo Clinic Rochester between 3/08/2007 and 12/8/2009. There were 13 cancelled participants and were excluded from baseline characteristics table.
Pre-assignment Details: Participants were evaluated by telephone, or in person, according to the eligibility criteria and educated about the requirements of the study. Eligible and willing women were registered onto the study.
Groups:
- Paced Breathing (15 Min Once Daily, 6 Breaths/Min): Patients practice paced breathing for 15 minutes once daily, 6 breaths/min, 5-7 days weekly, following an instructional compact disc (CD), for 8 weeks.
- Paced Breathing (15 Min Twice Daily, 6 Breaths/Min): Patients practice paced breathing for 15 minutes twice daily, 6 breaths/min, 5-7 days weekly, following an instructional compact disc (CD), for 8 weeks.
- Paced Breathing (10 Min Once Daily, 14 Breaths/Min): Patients practice paced breathing for 10 minutes once daily, 14 breaths/min, 5-7 days weekly, following an instructional compact disc (CD), for 8 weeks.
Period: Overall Study
Arm/Group | Paced Breathing (15 Min Once Daily, 6 Breaths/Min) | Paced Breathing (15 Min Twice Daily, 6 Breaths/Min) | Paced Breathing (10 Min Once Daily, 14 Breaths/Min)
Started | 30 | 31 | 31
Completed | 21 | 25 | 27
Not Completed | 9 | 6 | 4
Not completed — Withdrawal by Subject | 7 | 5 | 3
Not completed — Lost to Follow-up | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Paced Breathing (15 Min Once Daily, 6 Breaths/Min) | Paced Breathing (15 Min Twice Daily, 6 Breaths/Min) | Paced Breathing (10 Min Once Daily, 14 Breaths/Min) | Total
Number analyzed (Participants) | 30 | 31 | 31 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (8.4) | 54.4 (8.1) | 54.5 (8.7) | 53.4 (8.5)
Age, Customized [Number; unit: participants]
  Between 18 and 49 years | 15 | 8 | 9 | 32
  >=50 years | 15 | 23 | 22 | 60
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 31 | 31 | 92
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 30 | 31 | 31 | 92
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 31 | 31 | 92
Breast Cancer History [Number; unit: participants]
  Yes | 20 | 13 | 15 | 48
  No | 10 | 18 | 16 | 44
Average Frequency of Hot Flashes per day [Number; unit: participants]
  <4 Hot flashes per day | 1 | 2 | 6 | 9
  4-9 Hot flashes per day | 10 | 15 | 14 | 39
  >=10 Hot flashes per day | 19 | 14 | 11 | 44
Current tamoxifen, raloxifene, or aromatase inhibitor treatment [Number; unit: participants]
  Yes | 14 | 7 | 12 | 33
  No | 16 | 24 | 19 | 59

OUTCOME MEASURES:

1. Primary Outcome: The Difference in Hot Flash Score (Frequency and Severity) Between Baseline (Week 1) and Week 9
Description: Hot flash severity were graded from 1 to 4, as they range from mild, moderate, severe, or very severe. A hot flash score is defined by multiplying the daily frequency with the average hot flash severity. These scores are aggregated into average weekly hot flash activity scores for each patient.
Time Frame: Week 1 and Week 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paced Breathing (15 Min Once Daily, 6 Breaths/Min) | Paced Breathing (15 Min Twice Daily, 6 Breaths/Min) | Paced Breathing (10 Min Once Daily, 14 Breaths/Min)
Number analyzed (Participants) | 30 | 31 | 31
units on a scale | -6.5 (5.38) | -7.5 (8.14) | -6.5 (7.97)
Statistical Analysis 1: Comparison: Paced Breathing (15 Min Once Daily, 6 Breaths/Min) vs Paced Breathing (10 Min Once Daily, 14 Breaths/Min); Treatment effectiveness was measured using pairwise comparisons of hot flash score change from baseline in each paced breathing arm; Test type: Superiority or Other; p = 0.3679, Wilcoxon rank-sum
Statistical Analysis 2: Comparison: Paced Breathing (15 Min Twice Daily, 6 Breaths/Min) vs Paced Breathing (10 Min Once Daily, 14 Breaths/Min); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4715, Wilcoxon rank-sum

2. Secondary Outcome: Change From Baseline to Week 9 for PSQI Global Score
Description: The Pittsburgh Sleep Quality Index (PSQI) has 19 items and seven component scales: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep-wake disturbances, use of sleep medication, and daytime dysfunction. The scoring algorithm yields seven component scales on 0-3 scales which are summed to produce a global score on a 0-21 scale with higher values representing more severe sleep difficulty. The global score is translated into 0-100 scale with high values representing best quality of life (QOL). The habitual sleep efficiency component and global score was estimated using the worst-case scenarios for the values that were provided for PSQI question 4. Change from baseline to week 9 was calculated by subtracting the baseline scores from the scores at week 9.
Time Frame: Baseline and Week 9
Population: Includes all participants who completed both baseline and week 9 assessments.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Paced Breathing (15 Min Once Daily, 6 Breaths/Min) | Paced Breathing (15 Min Twice Daily, 6 Breaths/Min) | Paced Breathing (10 Min Once Daily, 14 Breaths/Min)
Number analyzed (Participants) | 17 | 22 | 18
units on a scale | 4.8 [-14.3 to 28.6] | 4.8 [-28.6 to 38.1] | 7.1 [-19.0 to 28.6]

3. Secondary Outcome: Change From Baseline to Week 9 on Blood Pressure Measurement
Description: Participants were taught home monitoring of blood pressure and provided with the sphygmomanometer. The measurements data were recorded on the Blood Pressure Measurement log. Change from baseline to week 9 was calculated by subtracting the baseline measurement from the measurement at week 9.
Time Frame: Baseline and Week 9
Population: Includes all participants who had both baseline and week 9 blood pressure measurements.
Measure: Median (Full Range); unit: mmHg
Arm/Group | Paced Breathing (15 Min Once Daily, 6 Breaths/Min) | Paced Breathing (15 Min Twice Daily, 6 Breaths/Min) | Paced Breathing (10 Min Once Daily, 14 Breaths/Min)
Number analyzed (Participants) | 19 | 24 | 25
mmHg
  Diastolic Blood Pressure Morning | -4.1 [-37.0 to 5.7] | -1.9 [-23.4 to 10.5] | -1.6 [-19.9 to 7.3]
  Diastolic Blood Pressure Evening | -2.1 [-10.5 to 3.7] | -1.7 [-7.6 to 7.5] | 0.5 [-15.6 to 7.3]
  Systolic Blood Pressure Morning | 1.0 [-14.0 to 9.4] | 0.1 [-55.2 to 19.6] | -0.4 [-14.2 to 17.6]
  Systolic Blood Pressure Evening | -0.6 [-16.2 to 10.6] | -3.4 [-14.2 to 14.3] | 2.2 [-16.6 to 11.7]

4. Secondary Outcome: Change From Baseline to Week 9 for POMS Total Score and Subscales
Description: Profile of Mood States (POMS) measures a variety of mood states including tension/anxiety, depression/dejection, anger/hostility, vigor/activity, fatigue/inertia and confusion/bewilderment. Each subscale consist of 5 items with a 5 points-scale (0=not at all, 1=a little, 2=moderately, 3=quite a bit and 4=extremely). The subscale scores were the sum of all five items. The total score was the sum of all subscale scores. The scores were then transformed into a 100-point scale with higher numbers indicating best quality of life (QOL). Change from baseline to week 9 was calculated by subtracting the baseline scores from the scores at week 9.
Time Frame: Baseline and Week 9
Population: Includes all participants who completed both baseline and week 9 assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paced Breathing (15 Min Once Daily, 6 Breaths/Min) | Paced Breathing (15 Min Twice Daily, 6 Breaths/Min) | Paced Breathing (10 Min Once Daily, 14 Breaths/Min)
Number analyzed (Participants) | 18 | 23 | 27
units on a scale
  POMS Total Score | 4.4 (9.2) | 5.2 (9.9) | 3.9 (13.1)
  Tension-Anxiety Subscale | 0 (16.0) | 5 (13.5) | 3 (20.7)
  Depression-Dejection Subscale | 1.1 (9.3) | 3.9 (13.2) | -0.6 (16.6)
  Confusion-Bewilderment Subscale | 5.6 (11.2) | 5.2 (9.7) | 0.9 (8.0)
  Fatigue-Inertia Subscale | 8.6 (19.0) | 12.4 (20.1) | 13.8 (23.3)
  Vigor-Activity Subscale | 8.1 (17.8) | 4.3 (21.5) | 4.6 (17.2)
  Anger-Hostility Subscale | 2.8 (14.5) | 0.5 (11.8) | 1.5 (18.8)

5. Secondary Outcome: Pearson Correlation Coefficients for Changes in Hot Flash Scores From Baseline to Week 9 With Changes in POMS Total Score and Subscales From Baseline to Week 9
Description: Profile of Mood States (POMS) measures a variety of mood states including tension/anxiety, depression/dejection, anger/hostility, vigor/activity, fatigue/inertia and confusion/bewilderment. Each subscale consist of 5 items with a 5 points-scale (0=not at all, 1=a little, 2=moderately, 3=quite a bit and 4=extremely). The subscale scores were the sum of all five items. The total score was the sum of all subscale scores. The scores were then transformed into a 100-point scale with higher numbers indicating best quality of life (QOL). Change from baseline to week 9 was calculated by subtracting the baseline scores from the scores at week 9. The correlation was estimated using Pearson correlation coefficients. The assessment of the Pearson Correlation Coefficients was the pre-specified Secondary outcome, and not the underlying changes in the POMS scores.
Time Frame: Baseline and Week 9
Population: Includes all participants who completed both baseline and week 9 assessments.
Measure: Number; unit: Correlation coefficient
Arm/Group | Paced Breathing (15 Min Once Daily, 6 Breaths/Min) | Paced Breathing (15 Min Twice Daily, 6 Breaths/Min) | Paced Breathing (10 Min Once Daily, 14 Breaths/Min)
Number analyzed (Participants) | 18 | 23 | 25
Correlation coefficient
  POMS Total Score | -0.05 | -0.32 | 0.29
  Tension-Anxiety Subscale | -0.18 | -0.36 | 0.19
  Depression-Dejection Subscale | -0.05 | -0.35 | 0.35
  Confusion-Bewilderment Subscale | 0.21 | -0.33 | 0.37
  Fatigue-Inertia Subscale | 0.32 | -0.20 | 0.26
  Vigor-Activity Subscale | -0.22 | 0.04 | 0.01
  Anger-Hostility Subscale | -0.25 | -0.25 | 0.21

6. Secondary Outcome: Change From Baseline to Week 9 for BFI Fatigue Scores
Description: Brief Fatigue Inventory (BFI) consist of 3 items that assess the severity of fatigue and 6 items that assess the impact of fatigue on daily functioning in a 10-points scale with 0 as no fatigue or does not interfere with daily functioning and 10 as bad fatigue or completely interferes. The scores for the six items were summed up to form a total interference score. The linear analogue scale of fatigue was a 10-points scale with 0 as no fatigue and 10 as bad fatigue. All scores were then transformed into 0 to 100 scale, with 100 as less fatigue/less interference. Change from baseline to week 9 was calculated by subtracting the baseline scores from the scores at week 9.
Time Frame: Baseline and Week 9
Population: Includes all participants who completed both baseline and week 9 assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paced Breathing (15 Min Once Daily, 6 Breaths/Min) | Paced Breathing (15 Min Twice Daily, 6 Breaths/Min) | Paced Breathing (10 Min Once Daily, 14 Breaths/Min)
Number analyzed (Participants) | 19 | 23 | 25
units on a scale
  Fatigue Right Now | 8.9 (25.8) | 13.5 (19.9) | 17.2 (28.8)
  Usual Fatigue: number analyzed (Participants) | 19 | 22 | 25
  Usual Fatigue | 16.3 (18.6) | 11.8 (18.9) | 12.4 (25.1)
  Worst Fatigue Last 24 Hours | 12.6 (32.8) | 18.7 (23.2) | 18.8 (33.1)

7. Secondary Outcome: Pearson Correlation Coefficients for Changes in Hot Flash Scores From Baseline to Week 9 With Changes in BFI Fatigue From Baseline to Week 9
Description: Brief Fatigue Inventory (BFI) consist of 3 items that assess the severity of fatigue and 6 items that assess the impact of fatigue on daily functioning in a 10-points scale with 0 as no fatigue or does not interfere with daily functioning and 10 as bad fatigue or completely interferes. The scores for the six items were summed up to form a total interference score. The linear analogue scale of fatigue was a 10-points scale with 0 as no fatigue and 10 as bad fatigue. All scores were then transformed into 0 to 100 scale, with 100 as less fatigue/less interference. Change from baseline to week 9 was calculated by subtracting the baseline scores from the scores at week 9. The correlation was estimated using Pearson correlation coefficients. The assessment of the Pearson Correlation Coefficients was the pre-specified Secondary outcome, and not the underlying changes in the BFI fatigue items scores.
Time Frame: Baseline and Week 9
Population: Includes all participants who completed both baseline and week 9 assessments.
Measure: Number; unit: Correlation coefficient
Arm/Group | Paced Breathing (15 Min Once Daily, 6 Breaths/Min) | Paced Breathing (15 Min Twice Daily, 6 Breaths/Min) | Paced Breathing (10 Min Once Daily, 14 Breaths/Min)
Number analyzed (Participants) | 19 | 23 | 23
Correlation coefficient
  Fatigue Right Now | -0.25 | -0.20 | -0.18
  Usual Fatigue: number analyzed (Participants) | 19 | 22 | 23
  Usual Fatigue | 0.13 | 0.06 | -0.12
  Worst Fatigue Last 24 hours | 0.11 | -0.36 | -0.11

8. Secondary Outcome: Change From Baseline to Week 9 for Symptom Distress Diary
Description: Symptom Experience Diary is a self-report diary of expected side effects from controlled breathing on 10-points scale with 10 represents symptoms all the time. Individual item scores were then transformed into 0 to 100 scale, with 100 indicates best quality of life (QOL). Change from baseline to week 9 was calculated by subtracting the baseline scores from the scores at week 9.
Time Frame: Baseline and Week 9
Population: Includes all participants who completed both baseline and week 9 assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paced Breathing (15 Min Once Daily, 6 Breaths/Min) | Paced Breathing (15 Min Twice Daily, 6 Breaths/Min) | Paced Breathing (10 Min Once Daily, 14 Breaths/Min)
Number analyzed (Participants) | 19 | 24 | 27
units on a scale
  Fatigue: number analyzed (Participants) | 19 | 24 | 25
  Fatigue | 15.3 (30.3) | 20.8 (21.0) | 17.2 (32.2)
  Abnormal Sweating: number analyzed (Participants) | 19 | 24 | 26
  Abnormal Sweating | 20.0 (41.8) | 24.6 (30.2) | 29.2 (41.1)
  Trouble Sleeping: number analyzed (Participants) | 18 | 23 | 27
  Trouble Sleeping | 18.3 (30.2) | 21.7 (28.2) | 11.9 (28.0)
  Nervousness: number analyzed (Participants) | 18 | 24 | 27
  Nervousness | 4.4 (22.3) | 4.2 (17.4) | 6.3 (27.9)
  Negative Mood: number analyzed (Participants) | 18 | 24 | 27
  Negative Mood | 6.1 (18.5) | 12.1 (24.0) | 7.8 (24.4)

9. Secondary Outcome: Pearson Correlation Coefficients for Changes in Hot Flash Scores From Baseline to Week 9 With Changes in Symptom Experience Diary From Baseline to Week 9
Description: Symptom Experience Diary is a self-report diary of expected side effects from controlled breathing on 10-points scale with 10 represents symptoms all the time. Individual item scores were then transformed into 0 to 100 scale, with 100 indicates best quality of life (QOL). Change from baseline to week 9 was calculated by subtracting the baseline scores from the scores at week 9. The correlation was estimated using Pearson correlation coefficients. The assessment of the Pearson Correlation Coefficients was the pre-specified Secondary outcome, and not the underlying changes in the Symptom Experience Diary item scores.
Time Frame: Baseline and Week 9
Population: Includes all participants who completed both baseline and week 9 assessments.
Measure: Number; unit: Correlation coefficient
Arm/Group | Paced Breathing (15 Min Once Daily, 6 Breaths/Min) | Paced Breathing (15 Min Twice Daily, 6 Breaths/Min) | Paced Breathing (10 Min Once Daily, 14 Breaths/Min)
Number analyzed (Participants) | 19 | 24 | 25
Correlation coefficient
  Fatigue: number analyzed (Participants) | 19 | 24 | 23
  Fatigue | -0.24 | 0.04 | 0.26
  Abnormal Sweating: number analyzed (Participants) | 19 | 24 | 24
  Abnormal Sweating | -0.43 | -0.30 | -0.20
  Trouble Sleeping: number analyzed (Participants) | 18 | 23 | 25
  Trouble Sleeping | -0.56 | -0.15 | -0.28
  Nervousness: number analyzed (Participants) | 18 | 24 | 25
  Nervousness | -0.30 | -0.43 | 0.15
  Negative Mood: number analyzed (Participants) | 18 | 24 | 25
  Negative Mood | -0.19 | 0.05 | 0.21

ADVERSE EVENTS:
Time Frame: Weekly during week 2 to week 9
Arm/Group | Paced Breathing (15 Min Once Daily, 6 Breaths/Min) | Paced Breathing (15 Min Twice Daily, 6 Breaths/Min) | Paced Breathing (10 Min Once Daily, 14 Breaths/Min)
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/31 | 0/31
Other Adverse Events (participants affected / at risk) | 5/30 | 7/31 | 2/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paced Breathing (15 Min Once Daily, 6 Breaths/Min) (N=30) | Paced Breathing (15 Min Twice Daily, 6 Breaths/Min) (N=31) | Paced Breathing (10 Min Once Daily, 14 Breaths/Min) (N=31)
Palpitations (Cardiac disorders) | 1 (1) | 2 (4) | 1 (1)
Influenza Symptoms (General disorders) | 0 (0) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 5 (10) | 4 (4) | 1 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes